CLINICAL TRIAL: NCT04573205
Title: Primary TBE Vaccination for the Elderly
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Anja Rosdahl, Principal Investigator, Region Örebro County
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: O2019-1
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tick-borne Encephalitis; Vaccine
Keywords: Elderly; Tick-borne Encephalitis; Vaccine
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — FSME-IMMUN vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- > 50 years (Experimental): Healthy individuals > 50 years of age divided into age groups 50-59 years, 60-69 years and >70 years, approximately 20 participants in each group.
  Vaccinated with 4 doses FSME immune Adult intramuscular injection according to the recommended primary vaccine Schedule in Sweden for individuals > 50 years of age, at time 0, 1, 2 and 7 months.
  Interventions: Drug: FSME-IMMUN Vaccine
- < 40 years (Active Comparator): Healthy individuals < 40 years of age. Vaccinated with 3 doses FSME immune Adult intramuscular injection according to the standard recommended primary vaccine at time 0, 1, and 7 months.
  Interventions: Drug: FSME-IMMUN Vaccine

INTERVENTIONS:
Drug: FSME-IMMUN Vaccine — 0.5 ml intramuscular injection scheduled in the two different arms

SUMMARY:
Tick-borne Encephalitis (TBE) can be prevented by vaccine. Vaccine failure, defined as a case of TBE regardless of previous vaccination, has been described and seems to be more predominant with increasing age, suggesting a less effective immune response following with increasing age. In fact previous studies has shown a reduced antibody response in elderly individuals compared to younger when vaccinated against TBE. As a result, in Sweden, an extra vaccine dose has been recommended during the primary vaccine schedule to individuals > 50 years of age. This alternative vaccine schedule has not been tested. The investigator aim to test if an extra vaccine dose in the primary vaccine schedule for those > 50 years of age improves the immune response and offers a corresponding immunity to younger individuals following TBE vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 50 years or between 18-40 years
* Man or woman
* God health
* Written informed consent

Exclusion Criteria:

* Previous vaccination against TBE
* Previous TBE infection
* Allergy or hypersensitivity to any substance in the vaccine
* Previously known or suspected infection with Japanese encephalitis, Dengue virus, West Nile fever or Yellow fever
* Information on previous vaccination against Yellow fever or Japanese encephalitis
* Acute illness, eg fever with malaise
* Immunosuppression, due to medication or disease
* Previous treatment with Rituximab or equivalent
* Autoimmune disease, including diabetes (diet or tablet-treated diabetes with good metabolic control is accepted, HbA1c < 6 %)
* Obesity, BMI > 40
* Moderate to severe renal failure including hemodialysis, estimated GFR < 30.
* Blood transfusion or immunoglobulins <3 months ago
* Pregnancy
* Any other illness where the investigator consider the subject unsuitable for the study
* The study subject does not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Serological response to vaccination with TBE vaccine following primary vaccination | NT measured 1 months after vaccination
  The proportion of individuals > 50 years that achieves protective levels following the extra primary vaccine dose compared to the proportion of individuals tha achieve protective levels of neutralizing antibodies following the second vaccine dose in those < 40 years.
Serological response to vaccination with TBE vaccine following the full vaccine scehdule | NT measured 1 months after vaccination
  The proportion of individuals > 50 years that achieves protective levels of neutralizing antibodies following the final primary schedule ( dose 4), compared to those < 40 years ( 3 doses).

SECONDARY OUTCOMES:
Cellular immunity in young and elderly ( immune cell expression) | Measured 7 days after vaccination
  T and B cell populations (flow cytometry) 7 days after TBE vaccination
Cellular immunity in young and elderly ( cytokine production) | Measured 7 days after vaccination
  Cytokine production ( Luminex) 7 days after TBE vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Region Örebro Län, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lindquist L, Vapalahti O. Tick-borne encephalitis. Lancet. 2008 May 31;371(9627):1861-71. doi: 10.1016/S0140-6736(08)60800-4. PMID 18514730
- [Background] Prymula R, Pollabauer EM, Pavlova BG, Low-Baselli A, Fritsch S, Angermayr R, Geisberger A, Barrett PN, Ehrlich HJ. Antibody persistence after two vaccinations with either FSME-IMMUN(R) Junior or ENCEPUR(R) Children followed by third vaccination with FSME-IMMUN(R) Junior. Hum Vaccin Immunother. 2012 Jun;8(6):736-42. doi: 10.4161/hv.20058. Epub 2012 Jun 1. PMID 22699436
- [Background] Jilkova E, Vejvalkova P, Stiborova I, Skorkovsky J, Kral V. Serological response to tick-borne encephalitis (TBE) vaccination in the elderly--results from an observational study. Expert Opin Biol Ther. 2009 Jul;9(7):797-803. doi: 10.1517/14712590903066711. PMID 19527104
- [Background] Hainz U, Jenewein B, Asch E, Pfeiffer KP, Berger P, Grubeck-Loebenstein B. Insufficient protection for healthy elderly adults by tetanus and TBE vaccines. Vaccine. 2005 May 9;23(25):3232-5. doi: 10.1016/j.vaccine.2005.01.085. PMID 15837226
- [Background] Hansson KE, Rosdahl A, Insulander M, Vene S, Lindquist L, Gredmark-Russ S, Askling HH. Tick-borne Encephalitis Vaccine Failures: A 10-year Retrospective Study Supporting the Rationale for Adding an Extra Priming Dose in Individuals Starting at Age 50 Years. Clin Infect Dis. 2020 Jan 2;70(2):245-251. doi: 10.1093/cid/ciz176. PMID 30843030
- [Background] Lindblom P, Wilhelmsson P, Fryland L, Matussek A, Haglund M, Sjowall J, Vene S, Nyman D, Forsberg P, Lindgren PE. Factors determining immunological response to vaccination against tick-borne encephalitis virus in older individuals. PLoS One. 2014 Jun 26;9(6):e100860. doi: 10.1371/journal.pone.0100860. eCollection 2014. PMID 24967619
- [Background] Stiasny K, Aberle JH, Keller M, Grubeck-Loebenstein B, Heinz FX. Age affects quantity but not quality of antibody responses after vaccination with an inactivated flavivirus vaccine against tick-borne encephalitis. PLoS One. 2012;7(3):e34145. doi: 10.1371/journal.pone.0034145. Epub 2012 Mar 26. PMID 22461903
- [Background] Weinberger B, Keller M, Fischer KH, Stiasny K, Neuner C, Heinz FX, Grubeck-Loebenstein B. Decreased antibody titers and booster responses in tick-borne encephalitis vaccinees aged 50-90 years. Vaccine. 2010 Apr 30;28(20):3511-5. doi: 10.1016/j.vaccine.2010.03.024. Epub 2010 Mar 21. PMID 20332047
- [Background] Askling HH, Rombo L, van Vollenhoven R, Hallen I, Thorner A, Nordin M, Herzog C, Kantele A. Hepatitis A vaccine for immunosuppressed patients with rheumatoid arthritis: a prospective, open-label, multi-centre study. Travel Med Infect Dis. 2014 Mar-Apr;12(2):134-42. doi: 10.1016/j.tmaid.2014.01.005. Epub 2014 Jan 29. PMID 24529746
- [Background] Wagner A, Garner-Spitzer E, Jasinska J, Kollaritsch H, Stiasny K, Kundi M, Wiedermann U. Age-related differences in humoral and cellular immune responses after primary immunisation: indications for stratified vaccination schedules. Sci Rep. 2018 Jun 29;8(1):9825. doi: 10.1038/s41598-018-28111-8. PMID 29959387
- [Background] Hopf S, Garner-Spitzer E, Hofer M, Kundi M, Wiedermann U. Comparable immune responsiveness but increased reactogenicity after subcutaneous versus intramuscular administration of tick borne encephalitis (TBE) vaccine. Vaccine. 2016 Apr 12;34(17):2027-34. doi: 10.1016/j.vaccine.2015.12.057. Epub 2016 Jan 6. PMID 26768126
- [Background] Garner-Spitzer E, Seidl-Friedrich C, Zwazl I, Hofer M, Kinaciyan T, Jarisch R, Stiasny K, Zlabinger GJ, Kundi M, Wiedermann U. Allergic patients with and without allergen-specific immunotherapy mount protective immune responses to tick-borne encephalitis vaccination in absence of enhanced side effects or propagation of their Th2 bias. Vaccine. 2018 May 11;36(20):2816-2824. doi: 10.1016/j.vaccine.2018.03.076. Epub 2018 Apr 16. PMID 29673942
- [Background] Garner-Spitzer E, Wagner A, Paulke-Korinek M, Kollaritsch H, Heinz FX, Redlberger-Fritz M, Stiasny K, Fischer GF, Kundi M, Wiedermann U. Tick-borne encephalitis (TBE) and hepatitis B nonresponders feature different immunologic mechanisms in response to TBE and influenza vaccination with involvement of regulatory T and B cells and IL-10. J Immunol. 2013 Sep 1;191(5):2426-36. doi: 10.4049/jimmunol.1300293. Epub 2013 Jul 19. PMID 23872054
- [Background] Svahn A, Linde A, Thorstensson R, Karlen K, Andersson L, Gaines H. Development and evaluation of a flow-cytometric assay of specific cell-mediated immune response in activated whole blood for the detection of cell-mediated immunity against varicella-zoster virus. J Immunol Methods. 2003 Jun 1;277(1-2):17-25. doi: 10.1016/s0022-1759(03)00111-x. PMID 12799036
- [Background] Eliasson H, Olcen P, Sjostedt A, Jurstrand M, Back E, Andersson S. Kinetics of the immune response associated with tularemia: comparison of an enzyme-linked immunosorbent assay, a tube agglutination test, and a novel whole-blood lymphocyte stimulation test. Clin Vaccine Immunol. 2008 Aug;15(8):1238-43. doi: 10.1128/CVI.00434-07. Epub 2008 Jun 18. PMID 18562568